CLINICAL TRIAL: NCT02764996
Title: An Exploratory Prospective Trial of Rescue Acupuncture for the Treatment of Acute Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWH20150084H
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture for Migraine (Experimental): Acupuncture treatments will be subject dependent, and points could include the N point (on scalp); various auricular points to include Shen Men, Point Zero, thalamus and Omega-2; body points to include Liver 2, Liver 3, Gall Bladder 20, bladder 10; and surface release over tense areas in the neck or shoulders
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
This will be an exploratory observational trial of rescue acupuncture for the treatment of acute migraine in military beneficiaries to gain information to inform the power analysis of a larger, more definitive trial. Researchers do not seek to definitively answer the question of whether this acupuncture protocol is effective; rather, we seek to estimate the proportion of migraine episodes that result in headache-free status 20-30 minutes, 2 hours, 4 hours, and 24 hours after an acupuncture treatment. Acupuncture treatments will be subject dependent, and points could include the N point (on scalp); various auricular points to include Shen Men, Point Zero, thalamus and Omega-2; body points to include Liver 2, Liver 3, Gall Bladder 20, bladder 10; and surface release over tense areas in the neck or shoulders. Researchers will document the points used, and data will be aggregated to determine overall effectiveness. Sub-group analysis by points will be performed to determine if there is more usefulness in 1 point or combination of points. These estimates will inform statistical power calculations for a future randomized controlled trial (RCT) that directly compares the effectiveness of Rescue Acupuncture with medical management of acute migraine with rescue medication. Researchers will also assess the feasibility of this study protocol as well as patient receptivity and satisfaction.

DETAILED DESCRIPTION:
Male and female (DoD beneficiaries). Age 18 years or older, who meet eligibility criteria will be offered an opportunity to participate via Primary Care Manager (PCM) referrals and posted advertisements will be utilized for recruiting subjects to the study. Some patients may be patients of the Principal Investigator or Associate Investigator, however, they will have the study staff recruit their patients to prevent any misconception of coercion or undue influence. When a potential subject is identified by the treating PCM, the patient will either be provide a contact number to the Research Staff, the Research Staff will be given the potential subjects contact information by the PCM, or the PCM will come and get the Research Staff to speak with the patient directly. Researchers will administer acupuncture treatments for up to 6 different migraine episodes per subject over the course of 3 months. This type of Acupuncture for this indication is routinely done as part of standard-of-care in our Family Medicine and acupuncture clinics both in conjunction with rescue medications and as a stand-alone therapy.

Screening Visit:

* Obtain signed Informed Consent document and HIPAA Authorization. (research only)
* Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria including previous encounter, vital signs review, medication list, co-morbidities, demographics, problems list, and note any prior acupuncture received. (research only)
* Record: Date of birth, age, gender, race, ethnicity, last 4 of social security number, name of standard of care rescue medications (over-the-counter and prescription), current email address (to be used for scheduling only), height (in inches), weight (in pounds), history of traumatic brain injury, concussion, or any mild to severe head trauma, medication use, history of acupuncture. (research only)
* Researchers will ask what the subjects expectations are regarding acupuncture's effectiveness for migraine. (research only)
* Researchers will instruct subjects not to take their over-the-counter and prescription headache medications until after their visit with the research staff. (Standard care)
* Researchers will instruct subjects to bring their over-the-counter and prescription headache medications with them to each visit if their symptoms do not resolve from the acupuncture treatment. (research only)
* Patient will be instructed to contact the Research Coordinator, as soon as possible, after onset of migraine symptoms (including prodromal symptoms) to schedule an emergent visit with the research staff. (research only)
* Patient will be given a contact card with the names and phone numbers of the research staff to contact when they have a migraine episode.

Migraine Episode:

* Self-reported headache pain severity (0=no headache, 1=mild, 2=moderate, 3=severe) (Standard care)
* Record type and amount of rescue medications (over-the-counter and prescription) use in the past 7 days. (research only)
* Acupuncture treatments will be subject dependent, and points could include the N point (on scalp); various auricular points to include Shen Men, Point Zero, thalamus and Omega-2; body points to include Liver 2, Liver 3, Gall Bladder 20, bladder 10; and surface release over tense areas in the neck or shoulders. (Standard care)
* Researchers will document the points used. (Standard care)

  *If after 20-30 minutes these patients have not had resolution of their headache, they may take their standard of care rescue medication. (research only)
* The subject will sit for 20-30 minutes post-acupuncture(research only), and then the needles will be removed and the subject will be asked:

  o Self-reported headache pain severity (0=no headache, 1=mild, 2=moderate, 3=severe) (research only)
* Subject is allowed to leave and will be informed of the following telephone follow ups:
* 2 Hours post acupuncture:

  o Self-reported headache pain severity (0=no headache, 1=mild, 2=moderate, 3=severe) (research only)
* 4 Hours post acupuncture:

  o Self-reported headache pain severity (0=no headache, 1=mild, 2=moderate, 3=severe) (research only)
* 24 Hours post acupuncture:

  * Self-reported headache pain severity (0=no headache, 1=mild, 2=moderate, 3=severe)
  * Would you use acupuncture for future pain management? (Yes or no)
  * Would you prefer acupuncture or your rescue meds (both over-the-counter and prescription) for future episodes?
  * Record type and amount of rescue medications (over-the-counter and prescription) used since acupuncture. (research only)

ELIGIBILITY:
Inclusion:

* Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study.
* Male and female DoD beneficiaries, age 18 years or older, who have been previously prescribed rescue medication to treat their acute migraine episodes.

Exclusion:

* Pregnant
* Absence of ear
* Active cellulitis of ear
* Ear anatomy precluding identification of acupuncture landmarks
* Use of Hearing Aids that preclude the insertion of needles
* Use of anticoagulants
* Unable to drive during rapid onset of migraine or inability to find someone to drive you

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bobnick, DO, Principal Investigator — Principal Investigator
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Researchers are not sharing data

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture for Migraine: Acupuncture treatments will be subject dependent, and points could include the N point (on scalp); various auricular points to include Shen Men, Point Zero, thalamus and Omega-2; body points to include Liver 2, Liver 3, Gall Bladder 20, bladder 10; and surface release over tense areas in the neck or shoulders
  Acupuncture
Period: Overall Study
Arm/Group | Acupuncture for Migraine
Started | 26
Completed | 18
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture for Migraine
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change of Migraine Headache Pain
Description: Change of migraine headache pain from mild, moderate or severe to pain free.
Time Frame: 24 hours post treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture for Migraine
Number analyzed (Participants) | 18
Participants
  Achieved pain free condition--yes | 16
  achieved pain free conditon--no | 2

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Acupuncture for Migraine
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02764996/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02764996/ICF_001.pdf